CLINICAL TRIAL: NCT00445068
Title: A Phase II Study Of Oral LBH589 In Adult Patients With Multiple Myeloma Who Have Received At Least Two Prior Lines Of Therapy And Whose Disease Is Refractory To The Most Recent Line Of Therapy
Brief Title: Efficacy and Safety of LBH589B in Adult Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2203
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; adults; LBH589; refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat

ARMS (1):
- Panobinostat (Experimental): Participants received panobinostat 20 milligrams (mg) orally once daily (OD), three times a week on days: 1, 3 and 5, then 8, 10 and 12, then 15, 17 and 19 of each cycle, as part of a 3-week (21 days) treatment cycle. Participants could continue treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat

SUMMARY:
This study will evaluate the efficacy and safety of LBH589B in adult patients with multiple myeloma who have received at least two prior therapies and are refractory to their last therapy. Patients must have received in prior therapy either bortezomib or lenalidomide

ELIGIBILITY:
Inclusion criteria:

1. Adults ≥ 18 years old
2. Subjects must have signed the consent form before undergoing any study specific screening procedures and before participation in this study. The subject must be fully informed by the investigator of the nature and potential risks of participation in this study.
3. Patients must have had a diagnosis of symptomatic multiple myeloma (from IMWG see (Kyle et al,2003) meeting all three of the following criteria:

   * Monoclonal immunoglobulin (spike on electrophoresis, or band on immunofixation) on serum or on 24 hour urine.
   * Bone marrow (clonal) plasma cells or plasmacytoma
   * Related organ or tissue impairment (anemia, hypercalcemia, lytic bone lesions, renal insufficiency, hyperviscosity or recurrent infections) (The Kyle et al 2003 definition of symptomatic Myeloma has been adapted based on the new exclusion criteria defined in protocol amendment 1)
4. Subjects must have received at least two prior lines of therapy and be refractory to the most recent line of therapy according to the following definitions: Refractory to most recent line of therapy Defined by disease progression during treatment or within 60 - 100 days after the completion of the most recent line of therapy. This includes the development of disease progression during maintenance or consolidation therapy with high dose glucocorticoids, or any other specific MM therapy Sixty days is counted from the point in time when the first response assessment is performed after completion of the last line of therapy. At a maximum, disease progression should be documented within 100 days after the last day of the last dose of any anti-MM therapy, including if last regimen of the most recent line of therapy was Autologous Stem Cell Transplant (ASCT). Stable disease patients also part of the IMWG definition are not eligible for this trial. At study screening, Progressive Disease (PD) will be assessed by comparing screening values or symptoms in reference to the baseline (values or symptoms) of their last line of therapy. Should a patient have experienced an initial response on their last line of therapy, PD should be assessed in reference to the lowest values of the initial confirmed response Minimal Response(MR) / Partial Response (PR) / Complete Response (CR).

   Disease progression is defined by having one or more of the following:
   * >25% increase in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation.
   * >25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200 mg/24 h and confirmed on a repeat investigation.
   * >25% increase in plasma cells in a bone marrow aspirate or on bone marrow biopsy, which must also be an absolute increase of at least 10%
   * Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas.
   * Development of new bone lesions or soft tissue plasmacytomas (not including compression fracture).
   * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.8 mmol/L not attributable to any other cause).
5. Subjects must have previously been treated with bortezomib and at least one of the following: lenalidomide or thalidomide
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
7. Patients must have the following hematological laboratory values:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L (or ≥1.0 x 109/L if the neutropenia is clinically related to progressive myeloma with bone marrow infiltration of > 50% involvement
   * Hemoglobin ≥ 8.0 g/dl
   * Platelets ≥ 75.0 x 109/L (or ≥ 50.0 x 109/L x if the thrombocytopenia is clinically related to progressive myeloma with bone marrow infiltration > 50% involvement
8. Patients must have the following renal function as shown by :

   * Calculated Creatinine Clearance (CrCL) > 30ml/min (Cockcroft and Gault formula)
9. Patients must have adequate liver function as shown by:

   * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 x Upper limit of normal (ULN)
   * Serum bilirubin ≤ 1.5 x ULN
   * Albumin ≥ 2.5 g/dl
10. Patients must have the following non-hematological laboratory values:

    * Serum potassium ≥ Lower Limit of Normal (LLN),
    * Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN,
    * Serum magnesium ≥ LLN
    * Serum phosphorus ≥ LLN
    * Normal thyroid function (TSH and free T4) (hypothyroidism correctable with supplements is allowed)
11. Baseline Multiple Uptake Gated Acquisition scan (MUGA) or echocardiogram (ECHO) must demonstrate Left Ventricular Ejection Fraction (LVEF) ≥ the lower limit of the institutional normal
12. Patients must be willing and able to undergo bone marrow aspirates as per protocol, with/without bone marrow biopsy according to their center's practice. The bone marrow aspirate /biopsy must be adequate to allow for comparison for the later efficacy response assessments.
13. Patients must have an M component at baseline above a minimum threshold of: 1g/dl (10g/L) for serum M component, or 200mg/24h urine M component.

Exclusion criteria:

1. Prior therapy with an Histone Deacetylase (HDAC) inhibitor for the treatment of Multiple Myeloma (MM)
2. Patients with non-secretory MM
3. Patients who have received allogenic stem cell transplantation < 12 months prior to study
4. Patients who have had prior allogenic stem cell transplantation and show evidence of active graft versus-host disease that requires immunosuppressive therapy
5. Patients with amyloidosis
6. Patients with peripheral neuropathy > grade 2
7. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Patients with congenital long QT syndrome
   * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as Heart Rate (HR)< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
   * Screening Electrocardiogram (ECG) with a corrected QT interval (QTc) > 450 msec
   * Right bundle branch block + left anterior hemi-block (bi-fascicular block)
   * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
8. Other clinically significant heart disease (e.g., Congestive Heart Failure (CHF NY) Heart Association class III or IV, uncontrolled hypertension, or history of poor compliance with an antihypertensive regimen)
9. Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
10. Patients with unresolved diarrhea > CTCAE grade 1.
11. Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
12. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsades de pointes if the medications cannot be discontinued or switched to a different medication prior to starting study drug
13. Concomitant use of CYP3A4 inhibitors
14. Patients with an active bleeding diathesis or on any treatment with therapeutic doses of sodium warfarin (Coumadin®) or any other anti-vitamin K drug. Low doses of Coumadin® (e.g., ≤ 2 mg/day), or low doses of any other anti-vitamin K drug, for line patency is allowable
15. Patients who have received chemotherapy, radiation therapy or any investigational drugs, bortezomib or other immunomodulatory therapy (e.g., thalidomide, lenalidomide) or immunotherapy ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such therapy
16. Patients who have received high-dose corticosteroids as the only component of their most recent line of therapy
17. Patients who have received steroids (e.g., dexamethasone) ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if subjects receive < 20 mg of prednisone or equivalent as indicated for other medical conditions (and not as maintenance or an anticancer therapy for MM), or up to 100 mg of hydrocortisone as premedication for a administration of certain medications or blood products, while enrolled in this study.
18. Patients whose clinical condition would need valproic acid therapy during study or ≤ 5 days prior to starting drug
19. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
20. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP)not willing to use a double method of contraception during the study and for 3 months after treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589
21. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and for 3 months after treatment. One of these methods of contraception must be a condom
22. Patients with a current second malignancy or a prior malignancy within the last 5 years except adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
23. Patients with any significant history of non compliance to medical regimens or unwilling or unable to comply with the protocol or unable to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-04-16 (Actual); Primary Completion 2008-05-19 (Actual); Study Completion 2009-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (24):
  - Mayo Clinic, Scottsdale, Arizona
  - Aptium Oncology, Berkeley, California
  - City of Hope, Duarte, California
  - UCSF, San Francisco, California
  - Stanford, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Christiana Care, Newark, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Dana Farber, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Hackensack University, Hackensack, New Jersey
  - Duke, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Metrohealth, Cleveland, Ohio
  - Sarah Canon Research Center, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - CTRC, San Antonio, Texas
- Germany (5):
  - Novartis investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Starnberg
  - Novartis Investigative Site, Würzburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in 6 countries
Pre-assignment Details: A total 38 participants were enrolled in the study, of which 38 discontinued the study.
Period: Overall Study
Arm/Group | Panobinostat
Started | 38
Completed | 2
Not Completed | 36
Not completed — Disease progression | 26
Not completed — Adverse Event | 5
Not completed — Abnormal laboratory value | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed Full Analysis Set (FAS) was defined according to the Intention to Treat (ITT) principle. This population included all participants enrolled into the study. Enrolled patients were those who had received at least one dose of study medication.
Groups:
- Panobinostat: Participants received panobinostat 20 mg orally OD, three times a week on days: 1, 3 and 5, then 8, 10 and 12, then 15, 17 and 19 of each cycle, as part of a 3-week (21 days) treatment cycle.
Arm/Group | Panobinostat
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5
  Caucasian | 31
  Other | 1
  Pacific islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response(CR) / Partial Response (PR))
Description: The response (complete response (CR) / partial response (PR)) rate as per Bladé criteria was assessed by the investigator. Response to treatment was evaluated in participants with multiple myeloma (MM) who have received at least two prior lines of therapy and whose disease was refractory to the most recent line of therapy.
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: The analysis was performed in Full Analysis Set (FAS) population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study. Enrolled patients were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated due to insufficient clinical efficacy in the targeted participants population. Due to insufficient data, this outcome could not be measured.
Groups:
- Panobinostat: Participants received panobinostat 20 mg orally OD, three times a week on days: 1, 3 and 5, then 8, 10 and 12, then 15, 17 and 19 of each cycle, as part of a 3-week (21 days) treatment cycle. Participants could continue treatment until disease progression or unacceptable toxicity.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is the proportion of patients with a best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria (Overall Response (OR) = CR + PR).
  Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study. Enrolled patients were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated due to insufficient clinical efficacy in the targeted participants population. Due to insufficient data, this outcome could not be measured.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined by the percentage of participants achieving either a confirmed tumor response or stable disease (SD) for at least 24 weeks. Response Criteria in Solid Tumors (RECIST) is a system for measuring tumor shrinkage or progression in terms of the longest dimensions of the tumor on imaging scans such as computerized tomography (CT). A "partial response" requires a decrease of 30% or more, "Progression" requires an increase of at least 20%, and "Stable disease" falls in between these two. All responses have a repeat assessment to confirm the response
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as time between time to first documented response (CR/PR) and time to first documented disease progression or death.
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response
Description: Time to response is defined as time between Day 1 cycle 1 and time to first documented response (CR/PR).
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressions free survival is defined as time between Day 1 cycle 1 and time to first documented disease progression or death. Disease progression will be determined as per response criteria.
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety and Tolerability
Description: Adverse Event (AE) are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: From Start of the Study up to 57 Weeks approximately.
Population: The analysis was performed on Safety population consisted of all participants who had received at least one dose of study medication and had one valid post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 38
Participants
  Participants with Adverse Events | 38
  Deaths | 7
  On treatment deaths | 3
  Serious Adverse Events | 17
  Study-drug-related Serious Adverse Events | 3
  Adverse Events Leading to discontinuation | 8

8. Secondary Outcome: Time to Peak Concentration (Tmax) of Panobinostat
Description: Tmax is defined as the time at which the Cmax occurs. It will be obtained from the Tmax parameter calculated by WinNonlin®. If there is no measurable Cmax in the subject's pharmacokinetic (PK) profile, then Tmax will be missing for that subject. Tmax will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in Pharmacokinetic Analysis (PAS) population, defined as all participants who provide at least one post-dose Pharmacokinetic (PK) plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Median (Full Range); unit: Hours
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Hours
  Day 1 | 1.7 [0.2 to 5.2]
  Day 8 | 1.2 [0.2 to 23.7]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Panobinostat
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations. It will be obtained from the Cmax parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Cmax will be missing for that subject. Cmax will be reported in units of ng/mL.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in PAS population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ng/mL
  Day 1 | 7.6 (5.52)
  Day 8 | 9.7 (6.51)

10. Secondary Outcome: Area Under the Plasma Concentration (AUC0-24) of Panobinostat
Description: Area under the curve (AUC) is defined as the area under concentration-time curve as a measure of drug exposure. The area under the plasma concentration-time curve from time zero to 24 hours.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ng*hr/ml
  Day 1 | 72.0 (36.10)
  Day 8 | 81.6 (37.56)

11. Secondary Outcome: Last Observed Plasma Concentration (Clast) of Panobinostat
Description: Clast is defined as the Last observed (quantifiable) plasma concentration (Clast), in units of ng/mL. Blood samples were collected to assess Clast.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ng/mL
  Day 1 | 0.3 (0.18)
  Day 8 | 1.1 (1.13)

12. Secondary Outcome: Time of Clast (Tlast) of Panobinostat
Description: Time of Clast (Tlast) will be obtained from the Tlast parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Tlast will be missing for that participants. Tlast will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Hours
  Day 1 | 47.8 [24 to 50.2]
  Day 8 | 24.3 [3.3 to 28.0]

ADVERSE EVENTS:
Time Frame: From Start of the Study up to 57 Weeks approximately.
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Arm/Group | Panobinostat
All-Cause Mortality (participants affected / at risk) | 7/38
Serious Adverse Events (participants affected / at risk) | 17/38
Other Adverse Events (participants affected / at risk) | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
General physical health deterioration (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Respiratory tract infection (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Monoclonal immunoglobulin present (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Uraemic encephalopathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Emotional distress (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=38)
Anaemia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 2
Fatigue (General disorders) | 18
Gait disturbance (General disorders) | 2
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 2
Pyrexia (General disorders) | 8
Gastrointestinal infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Blood creatinine increased (Investigations) | 10
Blood uric acid increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 4
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Renal failure acute (Renal and urinary disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes